CLINICAL TRIAL: NCT04081285
Title: Identification of Epigenetic Biomarkers for Alzheimer's Disease in Blood Using Epigenome-wide Analysis
Brief Title: Epigenetic Biomarkers for Alzheimer's Disease
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hong Kong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Timothy Kwok, Professor, Chinese University of Hong Kong
Other Study IDs: 2018.441
Record Dates: First submitted 2019-07-23; First posted 2019-09-09 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Alzheimer's disease (AD) is a neurodegenerative disorder with no know cure. The pathogenesis of late onset AD (LOAD) is complex and multifactorial in nature, with multiple susceptibility genes and environmental factors at interplay.

The objective of this study is to improve our understanding of the risk factors of LOAD by conducting an epigenome wide study within patients of LOAD contrasted against their cognitively normal siblings.

ELIGIBILITY:
Inclusion Criteria:

* Sufficient Cantonese competency for cognitive test
* Written informed consent given
* Have at least one gender-matched cognitively normal sibling

Exclusion Criteria:

* Subjects who refuse blood taking procedure
* Do not have a reliable family/caregiver informant (personal contact at least once a month)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Alzheimer's disease patients and normal siblings
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
DNA methylation | 5 years
RNA-seq microbiome | 5 years
Alzheimer's disease Assessment Scale-cognitive subscale (Adas-Cog) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Kwok, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong